CLINICAL TRIAL: NCT01874509
Title: Randomized Controlled Trial of a Minimal Versus Extended Internet-based Intervention for Problem Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFP 285651
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Alcohol Consumption; Hazardous Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Check Your Drinking screener (Active Comparator): Internet based program of lower intensity as compared to the "Alcohol Help Centre. It was designed to assesses drinking patterns, increase self-awareness of individual triggers, and set and achieve goals regarding abstinence.
  Interventions: Behavioral: Check Your Drinking
- Alcohol Help Centre (Experimental): Internet based program of higher intensity as compared to the "Check Your Drinking" intervention. It was designed to assesses drinking patterns, increase self-awareness of individual triggers, and set and achieve goals regarding abstinence.
  Interventions: Behavioral: Alcohol Help Centre

INTERVENTIONS:
Behavioral: Check Your Drinking
  Arms: Check Your Drinking screener
Behavioral: Alcohol Help Centre
  Arms: Alcohol Help Centre

SUMMARY:
Alcohol is one of the leading contributors to premature mortality and disability. Most people with alcohol problems will never seek treatment. There is a need to develop alternate ways to help problem drinkers outside of formal treatment settings.

One promising strategy is Internet-based interventions for problem drinkers. The first randomized controlled trial found that the investigators could reduce alcohol consumption by about six drinks per week at a six-month follow-up using a minimal, personalized feedback Internet-based intervention. The investigators second randomized trial demonstrated that an extended Internet-based intervention that contained a range of cognitive-behavioural and relapse prevention tools could produce greater reductions in problem drinking compared to that provided by the same minimal intervention at a six-month follow-up. Building upon this research, the current project will assess whether this extended Internet-based intervention can have a sustained impact on problem drinking. Specifically, the major objective of this project is to conduct a randomized controlled trial comparing the impact of an extended Internet-based self-help intervention for problem drinkers to a minimal Internet-based intervention in the general population of problem drinkers over a two year period.

Problem drinking participants will be recruited through media advertisements across Canada and will be randomly assigned to the minimal or extended Internet-based interventions. Six-month, twelve-month and two-year drinking outcomes will be compared between experimental conditions. It is predicted that participants receiving the extended Internet intervention will display sustained improved drinking outcomes compared to participants in the minimal Internet intervention condition. This programmatic line of research will advance the science of Internet-mediated intervention.

ELIGIBILITY:
Inclusion Criteria:•Resident of Canada

* 18 years of age or over
* A score of 8 or over on the Alcohol Use Disorders Identification Test (AUDIT)
* Indicate an interest in receiving self-help materials
* Have home access to the Internet
* Are willing to participate in follow-up at six month, twelve month and 2 year intervals

Exclusion Criteria:None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in AUDIT-C from baseline | 6 months, 1 year, 2 years
  A composite measure of three quantity/frequency drinking items (number of drinks per drinking day; frequency of alcohol consumption; frequency of 5+ drinking days). Developed by the world health organization.

SECONDARY OUTCOMES:
Change in number of drinks in a typical week from baseline | 6 months, 1 year, 2 years
  Sum of number of drinks consumed in a typical week
Change in highest number of drinks on one occasion from baseline | 6 months, 1 year, 2 years
  Greatest amount drunk on one occasion

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham JA, Shorter GW, Murphy M, Kushnir V, Rehm J, Hendershot CS. Randomized Controlled Trial of a Brief Versus Extended Internet Intervention for Problem Drinkers. Int J Behav Med. 2017 Oct;24(5):760-767. doi: 10.1007/s12529-016-9604-5. PMID 27770293
- [Derived] Cunningham JA, Hendershot CS, Rehm J. Randomized controlled trial of a minimal versus extended Internet-based intervention for problem drinkers: study protocol. BMC Public Health. 2015 Jan 21;15:21. doi: 10.1186/s12889-015-1347-8. PMID 25604206